CLINICAL TRIAL: NCT00862355
Title: Bioequivalence Study of SPARC147609 in Patients With Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DOX_2I_1476_09
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Ovarian Carcinoma
Keywords: Carcinoma; Ovary; Carcinoma Ovary
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): SPARC147609
  Interventions: Drug: SPARC147609
- 2 (Active Comparator): Reference147609
  Interventions: Drug: Reference147609

INTERVENTIONS:
Drug: SPARC147609 — IV infusion
  Arms: 1
Drug: Reference147609 — IV infusion
  Arms: 2

SUMMARY:
Bioequivalence study of SPARC147609

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting all of the following criteria will be considered for enrollment in the study:

  * Availability of subject for the entire study period and willingness to adhere to protocol requirements.
  * Patients with documented diagnosis of Ovarian Cancer and eligible for receiving a dose 50mg/m2 of Doxorubicin liposome(preferably on no other concomitant medication, however, if considered necessary, to be documented and given).
  * Patients at least 18-years of age or older. iv. Subjects who have no evidence of underlying disease (except ovarian cancer) during screening medical history and whose physical examination is performed within 21 days prior to commencement of the study.
  * Patients with Performance ≤ 2 on the ECOG performance scale. vi. Subjects whose screening laboratory values are within normal limits or considered by the clinical Investigator/Co-Investigator to be of no clinical significance.
  * Informed consent form given in written form.

Exclusion Criteria:

* History or presence of significant:

  * Allergy or Significant history of hypersensitivity or idiosyncratic reactions to Doxorubicin Hydrochloride and/or any related compounds etc.
  * Cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunologic, dermatologic, musculoskeletal, neurological or psychiatric disease.
  * Alcohol dependence, alcohol abuse or drug abuse or addiction with any recreational drug within past one year.
  * Clinically significant illness (except ovarian cancer)within 4 weeks before the start of the study v. Positive result to HIV, HCV, RPR and HBsAg.
  * Use of enzyme-modifying drugs (like Phenytoin, Carbamazepine, Barbiturates, Gresiofulvine etc.) in the previous 30 days before day 1 of this study and during the study.
* Donation of 350 mL or more of blood in the previous 90 days before day 1 of this study.
* Participation in another clinical trial within the preceding 90 days of study start
* Subjects who have:

  * Systolic blood pressure less than 90 mm of Hg or more than 140 mm of Hg
  * Diastolic blood pressure less than 60 mm of Hg or more than 90 mm of Hg
  * Pulse rate below 60/min. or above 100/min

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
90% confidence interval of the relative mean Cmax, AUC0-t, AUC0-∞, of the test and reference product | 2 cycles

SECONDARY OUTCOMES:
Treatment emergent adverse events | 2 cycles

CONTACTS AND LOCATIONS:
Locations (1):
- SPARC Site 1, Hyderabaad, Andhra Pradesh, India

REFERENCES:
- [Derived] Bhowmik S, Bhowmick S, Maiti K, Chakra A, Shahi P, Jain D, Rajamannar T. Two multicenter Phase I randomized trials to compare the bioequivalence and safety of a generic doxorubicin hydrochloride liposome injection with Doxil(R) or Caelyx(R) in advanced ovarian cancer. Cancer Chemother Pharmacol. 2018 Sep;82(3):521-532. doi: 10.1007/s00280-018-3643-3. Epub 2018 Jul 11. PMID 29995186